CLINICAL TRIAL: NCT03761043
Title: Fostering Engagement From Nurses in Promoting IV to PO Antimicrobial Conversion: The FERN-IPO Study
Brief Title: Nurse Promotion of IV to PO Antimicrobial Conversion
Acronym: FERN-IPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelowna General Hospital (Other Government)
Responsible Party: Principal Investigator, Sean Gorman, Pharmacy Coordinator, Clinical Quality & Research, Kelowna General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IH1803202
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Behavior Change; Bacterial Infections
Keywords: Nurse; Antibiotic step-down
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention Arm (No Intervention): The nurses will have not been exposed to the behavior change intervention.
- Post-Intervention Arm (Experimental): The nurses will have been exposed to the behavior change intervention.
  Interventions: Behavioral: Professional Behavior Change Intervention

INTERVENTIONS:
Behavioral: Professional Behavior Change Intervention — IV to PO antimicrobial conversion guidelines for nurses, nurse in-services and internet education sessions, IV to PO antimicrobial conversion health record reminder, endorsement from antimicrobial stewardship program, prescribers, and nurse educators.
  Other Names: Printed educational materials; Educational meetings; Educational outreach visits; Local opinion leaders; Reminders
  Arms: Post-Intervention Arm

SUMMARY:
This is a prospective, quasi-experimental, historically controlled study to evaluate if a behavioural change intervention informed by the COM-B model of behaviour change can improve nurses' self-perceived capability, opportunity, and motivation to engage in the assessment of patients who may be appropriate for IV to PO antimicrobial conversion. This study also seeks to determine if this translates into an increase in IV to PO antimicrobial conversion rates in the acute care setting.

DETAILED DESCRIPTION:
Current antimicrobial stewardship guidelines recommend appropriate and timely IV to PO antimicrobial conversion in hospitalized patients. Published rates of IV to PO antimicrobial conversion are consistently below 50% in eligible inpatients. Studies have suggested that nurses may be well positioned to provide a positive influence on prescriber behavior related to antimicrobial IV to PO conversion, however, no published research has evaluated the impact of nurses on antimicrobial IV to PO conversion rates. Published research has described the barriers and enablers to nurse participation in promoting antimicrobial IV to PO conversion using the COM-B model of behaviour change. This quasi-experimental study will evaluate whether determinants of nurse behaviour and their actual behaviour can be changed to increase antimicrobial IV to PO conversion rates in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Nineteen years of age or older
* Employed as a RN or LPN at KGH in any capacity (full-time, part-time or casual employee)
* Practicing on a medicine/thoracic surgery ward (4A) or medicine/oncology/respiratory ward (4B)

Exclusion Criteria:

* RNs or LPNs on orientation shifts/training
* RNs or LPNs not engaged in patient care
* Student nurses/nurses in training

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2019-04-07 (Actual)

PRIMARY OUTCOMES:
IV to PO antimicrobial conversion rate | Six months (three months pre-intervention, three months post-intervention)
  Incidence of IV to PO antimicrobial conversion (defined as the initiation of a PO antimicrobial within 24 hours of discontinuation of an IV antimicrobial during a single treatment course in a specific patient) before and after behavior change intervention

SECONDARY OUTCOMES:
Days of IV therapy prior to conversion to PO antimicrobial | Six months (three months pre-intervention, three months post-intervention)
  For treatment courses that undergo IV to PO antimicrobial conversion, the days of IV antimicrobial therapy prior to PO conversion before and after intervention
Nurse perceptions of capability, opportunity and motivation to promote IV to PO antimicrobial conversion | Six months (three months pre-intervention, three months post-intervention)
  Constructs are derived using the Theoretical Domains Framework and assess nurse perceived capability, motivation, and opportunity to promote IV to PO antimicrobial conversion using a 7-point Likert scale (1 - Strongly Disagree, 2 - Disagree, 3- Slightly Disagree, 4 - Neither Agree or Disagree, 5 - Slightly Agree, 6 - Agree, 7- Strongly Agree). The average Likert scale score for each of nine constructs (based on the Theoretical Domains Framework) will be calculated for the pre-intervention period and the post-intervention period. Change in the average Likert score for each construct (question) in the pre-intervention period versus the post-intervention period will be compared for each construct. A higher average Likert score on a construct in the post-intervention period compared to the pre-intervention period indicates improved perceptions about capability, opportunity, or motivation to promote IV to PO antimicrobial conversion.

OTHER OUTCOMES:
Balancing measure - Failed IV to PO antimicrobial conversion | Six months (three months pre-intervention, three months post-intervention
  Incidence of failed IV to PO antimicrobial conversion (defined as the re-initiation of an IV antimicrobial within seven days following IV to PO conversion of an antimicrobial during a single treatment course for a specific patient) pre and post-intervention
Subgroup Analysis 1: Nursing Unit Conversion Comparison | Six months (three months pre-intervention, three months post-intervention)
  Incidence of IV to PO antimicrobial conversion on nursing unit 1 (contains a clinical pharmacist) versus nursing unit 2 (does not contain a clinical pharmacist) pre and post-intervention
Subgroup Analysis 2: High Bioavailability Antimicrobial Conversion | Six months (three months pre-intervention, three months post-intervention)
  Incidence of IV to PO antimicrobial conversion for highly bioavailable (F ≥ 80%) antimicrobials pre and post-intervention
Subgroup Analysis 2: Non-High Bioavailability Antimicrobial Conversion | Six months (three months pre-intervention, three months post-intervention)
  Incidence of IV to PO antimicrobial conversion for non-highly bioavailable (F < 80%) antimicrobials pre and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Cox, PharmD, Principal Investigator — Interior Health Authority
Locations (1):
- Kelowna General Hospital, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher CC, Cox VC, Gorman SK, Lesko N, Holdsworth K, Delaney N, McKenna C. A theory-informed assessment of the barriers and facilitators to nurse-driven antimicrobial stewardship. Am J Infect Control. 2018 Dec;46(12):1365-1369. doi: 10.1016/j.ajic.2018.05.020. Epub 2018 Aug 1. PMID 30077436